CLINICAL TRIAL: NCT05552430
Title: Physical and Psychological Measures of Pain in Acute Orthopedic Injuries: Use of At-home Virtual Reality
Brief Title: Virtual Reality for Pain in Acute Orthopedic Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ryan A., Mace, PHD, Staff Psychologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P001500
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Injuries; Injury Arm; Injury;Sports; Injury, Knee; Injury Wrist; Injury, Ankle; Injury Foot; Injury, Hand; Injury Finger; Injury Leg
Keywords: pain; disability; injury; orthopedics; rehabilitation; mind-body
MeSH Terms: conditions — Wounds and Injuries; Arm Injuries; Athletic Injuries; Knee Injuries; Wrist Injuries; Ankle Injuries; Foot Injuries; Hand Injuries; Finger Injuries; Leg Injuries; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Skills-Based VR (Experimental): Participants will complete daily skills-based Virtual Reality (VR) sessions for 8 weeks (an average of 6 minutes per day) to determine the feasibility of at-home VR technology to aid the recovery of acute orthopedic musculoskeletal injuries. The VR device software is equipped with pain-specific treatment modules (e.g., Pain Education, Relaxation/Interoception, Mindful Escapes, and Pain Distraction Games) derived from evidence-based principles of cognitive behavioral therapy (CBT), mindfulness, and pain neuroscience education.
  Interventions: Device: RelieveVRx

INTERVENTIONS:
Device: RelieveVRx — Participants will complete daily skills-based Virtual Reality (VR) sessions for 8 weeks (an average of 6 minutes per day) to determine the feasibility of at-home VR technology to aid the recovery of acute orthopedic musculoskeletal injuries. The VR device software is equipped with pain-specific treatment modules (e.g., Pain Education, Relaxation/Interoception, Mindful Escapes, and Pain Distraction Games) derived from evidence-based principles of cognitive behavioral therapy (CBT), mindfulness, and pain neuroscience education.

SUMMARY:
The goal of this study is to pilot test a skills-based virtual reality (VR) for acute orthopedic injury. It will measure the feasibility, signals of improvement, exploratory pain mechanisms, and user experience of an established skills-based program (RelieveVRx) for acute orthopedic injury.

DETAILED DESCRIPTION:
This study will use mixed-methods to investigate the feasibility of skills-based virtual reality (VR) for acute orthopedic injury in an open pilot with individual exit interviews (target N=10). Participants will be patients with acute orthopedic musculoskeletal injuries who are at risk for chronic pain and disability (PCS ≥ 20 and PASS-20 ≥ 40) and meet inclusionary/exclusionary criteria. Participants will be recruited through the MGH Orthopedics Department, flyers, and the Rally research platform. Participants will self-administer a skills-based virtual reality (VR) program at home over an 8-week period. Participants will attend two in-person study assessments to complete study assessments (surveys and an fNIRS imaging session). The primary outcome for the pilot will be a-priori Go/No-Go feasibility markers (feasibility, acceptability, fidelity, credibility, expectancy, satisfaction) of the VR program and data collection procedures to increase the success of subsequent trials. Exploratory measures include: multi-modal assessment of pain intensity, pain-specific coping (catastrophizing, self-efficacy, acceptance), disability, physical function, and emotional function (depression, anxiety, stress). The VR headset will collect usage data and daily smartphone surveys will track changes in pain during the 8-week intervention. Completers will have the opportunity to attend 30 min individual exit interviews to understand patients' perception of the VR and their experience with the study procedures to increase the success of larger trials.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient adults in the Level 1 Trauma Center
2. Age 18 or older
3. Able to meaningfully participate meaningfully (English fluency and literacy) and stable living situation
4. Acute musculoskeletal injury (e.g., fracture, dislocation, rupture) 1-2 months earlier (acute phase).
5. Pain Catastrophizing Scale ≥20 or Pain Anxiety Symptom Scale-20 ≥40
6. Has access to internet (Wi-Fi or wireless)
7. Willing to participate and comply with the requirements of the study protocol, including virtual reality program and questionnaire completion No psychotropics or stable for >6 weeks
8. Free of concurrent psychotropic medication for at least 2 weeks prior to initiation of treatment, OR stable on current psychotropic medication for a minimum of 6 weeks and willing to maintain a stable dose (i.e., no psychotropics or stable for >6 weeks)
9. Cleared by orthopedic surgeon for study participation

Exclusion Criteria:

1. Current or prior diagnosis of epilepsy, seizure disorder, dementia, migraines, or other neurological diseases that are contraindicated for VR
2. Medical condition predisposing to nausea or dizziness.
3. Hypersensitivity to flashing light or motion.
4. Vision or severe hearing impairment.
5. Injury to eyes, face, or neck that impedes comfortable use of virtual reality
6. Diagnosed with a medical illness expected to worsen in the next 3 months (e.g., malignancy)
7. Other serious injuries that occurred with the orthopedic injury or surgical complications (e.g., infection, need for repeat surgery)
8. Current or prior untreated mental illness, substance use disorder, or suicidal ideation
9. Self-reported pregnancy
10. Currently in litigation or under Workman's Comp
11. Practice of cognitive-behavioral therapy, yoga/meditation, or other mind body techniques once per week for 45 minutes or more within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan A Mace, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No enrolled participants were excluded from the study.
Period: Overall Study
Arm/Group | Skills-Based VR
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Marital Status [Count of Participants; unit: Participants]
  Married | 3
  Single, never married | 5
  Separated or Divorced | 1
  Widowed | 1
Education [Count of Participants; unit: Participants]
  Some college/Associates degree (<16 years) | 1
  Completed college (16 years) | 3
  Graduate/professional degree (>16 years) | 6
Employment [Count of Participants; unit: Participants]
  Employed full-time | 8
  Employed part-time | 1
  Unemployed | 1
Income [Count of Participants; unit: Participants]
  $15,000 to less than $20,000 | 1
  $50,000 to less than $75,000 | 3
  $75,000 or more | 6

OUTCOME MEASURES:

1. Primary Outcome: Credibility and Expectancy Questionnaire (CEQ)- Credibility Subscale
Description: Participants' perceived credibility, determined by the percentage of participants with scores (range = 3-27, higher scores mean better outcomes) over the scale's midpoint (≥70% good, ≥ 80% excellent).
Time Frame: Pre-intervention (week 0) only
Measure: Count of Participants; unit: Participants
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Participants | 8

2. Primary Outcome: Credibility and Expectancy Questionnaire (CEQ)- Expectancy Subscale
Description: Participants' treatment expectancy, determined by the percentage of participants with scores (range = 3-27, higher scores mean better outcomes) over the scale's midpoint (≥70% good, ≥ 80% excellent).
Time Frame: Pre-intervention (week 0) only
Measure: Count of Participants; unit: Participants
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Participants | 9

3. Primary Outcome: Client Satisfaction Questionnaire
Description: Participants' treatment satisfaction, determined by the percentage of participants with scores (range = 3-12) over the scale's midpoint (≥70% good, ≥ 80% excellent).
Time Frame: Post-intervention (week 8) only
Measure: Count of Participants; unit: Participants
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Participants | 9

4. Primary Outcome: System Usability Scale
Description: Assess global user experience of the VR device, with higher percentile rankings (range = 0-100) indicating greater usability. Usability was determined by the number of participants with System Usability Scale scores 68 and above (≥70% good, ≥ 80% excellent).
Time Frame: Post-intervention (week 8) only
Measure: Count of Participants; unit: Participants
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Participants | 8

5. Secondary Outcome: Patient's Global Impression of Change
Description: The number of participants that improved "much or very much" or "minimally" on the Patient's Global Impression of Change Scores for pain, emotional, and physical function during the VR program.
Time Frame: Post-intervention (week 8) only
Measure: Count of Participants; unit: Participants
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Participants | 10

6. Secondary Outcome: Motion Sickness and Nausea
Description: Assess adverse experiences with VR, determined by the percentage of participants with responses (range = 0 never to 3 always) below the scale's midpoint (≥70% good, ≥ 80% excellent).
Time Frame: Post-intervention (week 8) only
Measure: Count of Participants; unit: Participants
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Participants | 10

7. Secondary Outcome: Feasibility of Enrollment
Description: We will report the number of participants who agree to participate out of those eligible, evaluated at the end of study for all participants (≥70% good, ≥ 80% excellent).
Time Frame: Throughout the study completion, approximately 1 year
Population: This benchmark indicates the number of participants enrolled out of total eligible. More participants were deemed eligible than the number that enrolled, ultimately making the overall number of participants greater than the number stated in the participant flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 12
Participants | 10

8. Secondary Outcome: Acceptability of Treatment
Description: Acceptability of treatment was determined by the percentage of participants who completed at least 6 of 8 weeks of VR modules (≥70%, good; ≥ 80% excellent).
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Count of Participants; unit: Participants
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Participants | 10

9. Secondary Outcome: Adherence to Pain Surveys
Description: Adherence to Pain Surveys was determined by the percentage of participants who responded to at least 5/7 days for at least 6/8 weeks during the intervention period (≥70% good, ≥80% excellent).
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Count of Participants; unit: Participants
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Participants | 8

10. Secondary Outcome: Feasibility of Outcome Assessments
Description: The feasibility of data collection was determined by the percentage of participants with no missing outcomes data (≥70% good, ≥80% excellent).
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Count of Participants; unit: Participants
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Participants | 10

11. Other Pre Specified Outcome: Non-narcotic Pain Medications
Description: Number of days that non-narcotic pain medications were taken in the last week.
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Population: Out of 10 total participants, only 6 were included in the analysis for the Outcome Measure as they were taking non-narcotic medications during the study.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 6
days per week
  Pre-intervention | 1.9 (2.23)
  Post-intervention | 0.6 (0.97)

12. Other Pre Specified Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance
Description: The PROMIS Sleep Disturbance is an 8-item self-report of challenges affecting sleep and overall sleep quality and satisfaction over the past seven days. PROMIS Sleep Disturbance items are scored between 1 and 5: not at all (1) to very much (5), never (1) to always (5), and very poor (1) to very good (5). Total raw scores are converted to T-scores, with higher T-score values (e.g., 50 indicates the population mean with a standard deviation of 10) indicating worse outcome (greater sleep disturbance or worse sleep quality).
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
T-score
  Pre-intervention | 57.86 (7.94)
  Post-intervention | 47.27 (9.55)

13. Other Pre Specified Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function
Description: The PROMIS Physical Function is an 8-item self-report to assess participants' general ability to complete daily living activities. PROMIS Physical Function items are scored on a 1 (unable to do) to 5 (without any difficulty) or 1 (cannot do) to 5 (not at all) point scale. Total scores are converted to T-scores, with higher T-score values (e.g., 50 indicates the population mean with a standard deviation of 10) indicating greater better outcome (higher physical function).
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
T-score
  Pre-intervention | 35.32 (6.86)
  Post-intervention | 43.26 (7.13)

14. Other Pre Specified Outcome: Short Musculoskeletal Functional Assessment (SMFA) Questionnaire- Dysfunction Index
Description: The Short Musculoskeletal Function Assessment (SMFA) is a 46-item self-report to assess the extent to which one's injury interferes with their ability to complete daily living activities. The SMFA Dysfunction Intex contains 34 items that assess musculoskeletal function. SMFA items are scored on a 1 (no problems/difficulty) to 5 (unable to do) scale. Total scores are calcuted by summing items 1-34 for the Dysfunction Index. Total scores are standardized [(Actual raw score - lowest possible raw score/possible raw score range) *100], with high scores indicating poor function (standardized subscale range, min = 0, max = 100).
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Mean (Standard Deviation); unit: Standardized subscale score
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Standardized subscale score
  Pre-intervention | 51.93 (8.45)
  Post-intervention | 35.46 (7.59)

15. Other Pre Specified Outcome: Short Musculoskeletal Functional Assessment (SMFA) Questionnaire - Bother Index
Description: The Short Musculoskeletal Function Assessment (SMFA) is a 46-item self-report to assess the extent to which one's injury interferes with their ability to complete daily living activities. The SMFA Bother Index has 12 items that assess symptom burden. SMFA items are scored on a 1 (no problems/difficulty) to 5 (unable to do) scale. Total scores are calculated by summing items 35-46 for the Bothersome Index. Total scores are standardized [(Actual raw score - lowest possible raw score/possible raw score range) *100], with high scores indicating poor function (standardized subscale range, min = 0, max = 100).
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Mean (Standard Deviation); unit: Standardized subscale score
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
Standardized subscale score
  Pre-intervention | 60.76 (10.61)
  Post-intervention | 38.17 (11.18)

16. Other Pre Specified Outcome: Numerical Rating Scale (NRS) - Pain at Rest
Description: The Numerical Rating Scale (NRS) is a 2-item self-report that assesses participants' pain intensity at rest during the past week. One of two NRS items (pain at rest) is reported and scored on a 0 (no pain) to 10 (worst ever) scale.
Time Frame: Assessed Pre-intervention (week 0), Bi-weekly, Post-intervention (week 8). Pre-intervention (week 0) and Post-intervention (week 8) reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 3.50 (1.27)
  Post-intervention | 1.00 (0.94)

17. Other Pre Specified Outcome: Numerical Rating Scale (NRS) - Pain With Activity
Description: The Numerical Rating Scale (NRS) is a 2-item self-report that assesses participants' pain intensity with activity during the past week. One of two NRS items (pain with activity) reported and scored on a 0 (no pain) to 10 (worst ever) scale.
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 6.30 (1.64)
  Post-intervention | 2.90 (1.79)

18. Other Pre Specified Outcome: Pain Catastrophizing Scale (PCS)
Description: The Pain Catastrophizing Scale (PCS) is a 13-item self-report of catastrophic thoughts and emotions related to pain. The PCS-13 is scored on 0 (not at all) to 4 (all the time) scale. Higher scores (range = 0-52) indicate greater pain catastrophizing.
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 23.90 (9.62)
  Post-intervention | 7.50 (5.08)

19. Other Pre Specified Outcome: Pain Anxiety Scale (PASS)
Description: The Pain Anxiety Symptoms Scale (PASS) is a 20-item self-report of fear and anxiety related to pain. The PASS-20 is scored on 0 (never) to 5 (always) scale. Higher scores (range= 0-100) indicate greater pain anxiety.
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 51.10 (17.40)
  Post-intervention | 18.40 (12.80)

20. Other Pre Specified Outcome: Pain Self-Efficacy Questionnaire (PSEQ)
Description: The Pain Self-Efficacy Questionnaire is a 10-item self-report that measures participants' confidence in completing daily tasks and leisure activities despite experiencing pain. PSEQ items are scored on a 0 (not at all confident) to 6 (completely confident) scale. Higher total sum scores (total range = 0-60) indicate greater better outcome (pain self-efficacy).
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 35.50 (12.67)
  Post-intervention | 50.90 (6.95)

21. Other Pre Specified Outcome: Center for Epidemiologic Study of Depression (CESD) Scale
Description: The Center for Epidemiological Studies Depression Scale (CES-D) is a 20-item self-report that assesses how often participants' experience symptoms of depression in the last week. CES-D items are scored on a 0 (rarely or none of the time, less than 1 day) to 3 (most or all of the time, 5-7 days) scale. Higher scores (range = 0-60) indicate greater depressive symptoms.
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 20.00 (8.63)
  Post-intervention | 10.90 (6.61)

22. Other Pre Specified Outcome: Cognitive and Affective Mindfulness Scale (CAMS)
Description: The Cognitive and Affective Mindfulness Scale - Revised (CAMS-R) is a 12-item self-report that measures mindfulness principles: attention regulation, present focus, awareness, and non-judgmental awareness. CAMS-R items are scored on a 1 (rarely/not at all) to 4 (almost always) scale. Higher total scores (range = 12-48) indicate greater use of mindfulness.
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 31.20 (3.88)
  Post-intervention | 35.90 (5.92)

23. Other Pre Specified Outcome: Defense and Veterans Pain Rating Scale (DVPRS) - Activity Subscale
Description: The Defense and Veterans Pain Rating Scale (DVPRS) is a 4-item self-report that measures the extent to which pain interferes with usual activity, sleep, mood, and stress. One of four DVPRS (Activity Subscale) reported and scored on 0 (does not interfere) to 10 (completely interferes) scale.
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 6.90 (2.56)
  Post-intervention | 2.00 (2.05)

24. Other Pre Specified Outcome: Defense and Veterans Pain Rating Scale (DVPRS) - Sleep Subscale
Description: The Defense and Veterans Pain Rating Scale (DVPRS) is a 4-item self-report that measures the extent to which pain interferes with usual activity, sleep, mood, and stress. One of four DVPRS (Sleep Subscale) reported and scored on 0 (does not interfere) to 10 (completely interferes) scale.
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 5.90 (3.41)
  Post-intervention | 1.80 (2.74)

25. Other Pre Specified Outcome: Defense and Veterans Pain Rating Scale (DVPRS) - Mood Subscale
Description: The Defense and Veterans Pain Rating Scale (DVPRS) is a 4-item self-report that measures the extent to which pain interferes with usual activity, sleep, mood, and stress. One of four DVPRS (Mood Subscale) reported and scored on 0 (does not interfere) to 10 (completely interferes) scale.
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 6.00 (1.83)
  Post-intervention | 2.10 (1.79)

26. Other Pre Specified Outcome: Defense and Veterans Pain Rating Scale (DVPRS) - Stress Subscale
Description: The Defense and Veterans Pain Rating Scale (DVPRS) is a 4-item self-report that measures the extent to which pain interferes with usual activity, sleep, mood, and stress. One of four DVPRS (Stress Subscale) reported and scored is scored on 0 (does not interfere) to 10 (completely interferes) scale.
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 6.40 (1.51)
  Post-intervention | 2.20 (2.10)

27. Other Pre Specified Outcome: Measure of Current Status (MOCS)
Description: The Measure of Current Status (MOCS) is a 13-item self-report of the ability to use various skills to cope with daily stressors. MOCS items are scored on a 0 (I cannot do this at all) to 4 (I can do this extremely well) scale. Higher total scores (range = 0-52) indicate greater ability and confidence to utilize coping skills.
Time Frame: Pre-intervention (week 0), Post-intervention (week 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills-Based VR
Number analyzed (Participants) | 10
score on a scale
  Pre-intervention | 2.19 (0.53)
  Post-intervention | 2.78 (0.64)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between baseline (Week 0) and post-test assessments (Week 9).
Arm/Group | Skills-Based VR
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Skills-Based VR (N=10)
Brief, unrelated hospitalization (Infections and infestations) | 1 (1) — ID 3 reported a 3-day inpatient hospitalization for a hip cyst unrelated to the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Skills-Based VR (N=10)
Mild, related event due to "scuba" module (Psychiatric disorders) | 1 (1) — ID 4 discontinued module 22 because they were "startled" by unexpectedly seeing a scuba diver in the immersive underwater environment. This was deemed a mild adverse event that was resolved by the participant skipping the module.
fNIRS Movement (Psychiatric disorders) | 1 (1) — RA observed ID8 becoming tearful while moving their injured limb during visit. RA assessed discomfort, and ID8 requested to proceed with protocol. ID8 did not display further signs of discomfort and confirmed interest in continuing the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT05552430/Prot_SAP_000.pdf